CLINICAL TRIAL: NCT04603963
Title: Efects of Inspiratory Muscle Training in Patients With COVID-19 After Acute Phase. Prospective Study
Brief Title: Inspiratory Muscle Training in Patients With COVID-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was a change in the institutional flow reducing the cases of covid 19
Sponsor: Elaine Cristina Pereira <elaine.cpereira@einstein.br> (Other)
Responsible Party: Sponsor-Investigator, Elaine Cristina Pereira <elaine.cpereira@einstein.br>, physiotherapist, Hospital Israelita Albert Einstein
Organization: Hospital Israelita Albert Einstein (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34931220.1.0000.0071
Record Dates: First submitted 2020-10-25; First posted 2020-10-27 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Respiratory Disease
Keywords: physiotherapy; exercises; respiratory muscle training
MeSH Terms: conditions — COVID-19; Respiration Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Only patients with respiratory muscle weakness that were considered as the maximum inspiratory pressure value (less than or equal to 60% of the predicted value) entered for randomization. Stratified randomization was performed in which the impaired chest tomography (absent, less than 50% or greater than 50%) was taken into account to be randomly allocated to the groups.
Who Masked: Investigator
Masking Description: Stratified randomization was performed in which the impaired chest tomography (absent, less than 50% or greater than 50%)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group control (No Intervention): alternate exercises: in one day breathing exercises, active or with a load of large muscle groups (according to tolerance) with a maximum limit of 2 kg, sedation out of bed, walking. On another day aerobic exercise with cycle ergometer limited to 30 minutes.
- intervention group (Experimental): He received the same intervention as the control group, associating respiratory muscle training 1 time a day with power breathe 3 series of 10 repetitions (started with 30% of the Pimax value) with readjusted load every 7 days.
  Interventions: Device: power breathe

INTERVENTIONS:
Device: power breathe — respiratory muscle training 1 time a day with power breathe 3 sets of 10 repetitions
  Arms: intervention group

SUMMARY:
COVID 19 has become a pandemic and has led to high demand on healthcare systems. It can cause a severe acute respiratory syndrome (SARS CoV-2) which leads to a long hospital stay, developing important functional damage and making hospital discharge difficult. Elderly, obese and people with chronic diseases are more susceptible to contracting the disease, this profile of patients already has a predisposition for respiratory muscle weakness and in this context, after clinical stability, it is still necessary in a hospital environment to approach respiratory and motor physiotherapy. to optimize the recovery of these patients. Objective: Improved breathing, functionality, exercise capacity and muscle strength in non-critical patients. Method: Prospective randomized clinical study where one group received motor and respiratory physiotherapy and the other group performed the same therapy associated with inspiratory muscle training. Results: The findings will be compared before and after the approach and will be presented in graphs and tables. Statistical tests will be used considering a significance level of 5%.

DETAILED DESCRIPTION:
Prospective clinical study in patients with COVID-19 admitted to a non-critical unit of a tertiary hospital. They were randomized into a group that received motor and respiratory exercises and another group that received the same exercises associated with respiratory muscle training.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with COVID-19 through PCR aged over 18 years admitted to non-critical units.

Exclusion Criteria:

* patients with changes in the level of consciousness and non-transient understanding, exclusive palliative care without prognosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
impact on functionality | 14 days
  respiratory muscle training appears to impact functionality

CONTACTS AND LOCATIONS:
Locations (1):
- Municipal Hospital Vila Santa Catarina, São Paulo, Brazil